CLINICAL TRIAL: NCT02112604
Title: Determining Predictors of Adequate Upper Airway Function in Ventilated Patients
Brief Title: Predictors of Upper Airway Function and Sleep-disordered Breathing in the Critically Ill
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Director of Research, Critical Care Division; Associate Professor of Anaesthesia, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2010P001919B
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Critically Ill; Obstructive Sleep Apnea
Keywords: critically ill, OSA, mechanical ventilation
MeSH Terms: conditions — Critical Illness; Sleep Apnea, Obstructive | interventions — Ventilators, Mechanical; Respiratory Physiological Phenomena; Hypnotics and Sedatives

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ventilated patients: Patients who have been extubated within 24 hours and have been mechanically ventilated for at least 24 hours. Alice PDx, pulmonary function tests, muscle strength tests, grip strength measurements, ventilator, Sedatives and muscle relaxants given in the ICU
  Interventions: Device: Ventilator; Device: Alice PDx; Other: Pulmonary function test; Other: Muscle strength tests; Other: Grip strength measurement; Drug: Sedatives and muscle relaxants given in the ICU

INTERVENTIONS:
Device: Ventilator — Mechanical ventilator used to replace or assist spontaneous breathing.
Device: Alice PDx — Alice PDx is a polysomnography monitor used to study stages of sleep and detect sleep-disordered breathing. The device monitors PO2, airflow, EEG, EOG and abdominal wall movements to detect sleep apnea.
Other: Pulmonary function test — The pulmonary function tests are used to study upper airway patency.
Other: Muscle strength tests — MRC score (0-60) is a clinical assessment of muscle power on abduction of the arm, flexion of the forearm, extension of the wrist, flexion of the leg, extension of the knee and dorsal flexion of the foot with the score of (0-5) on each measurement
Other: Grip strength measurement — Grip strength has been shown to be an accurate means of assessing muscle function in the critically ill. Muscle weakness may have an impact on upper airway patency.
Drug: Sedatives and muscle relaxants given in the ICU — Patients in the ICU are administered sedatives, anesthetics, opiods, anti-pyschotics and neuromuscular blocking agents as part of routine care. We hypothesize that the use of these drugs is associated with sleep-disordered breathing following extubation. We will collect the drug doses from the patient's chart.

SUMMARY:
This is part 2 of the #NCT01618240 under the same IRB protocol #2010P001919. The primary objective of this study is to examine factors that are related to sleep-disordered breathing and upper airway patency in critically ill patients who have been recently mechanically ventilated. Our primary hypothesize is that sedatives and neuromuscular blocking agents given in the ICU prior to extubation and during the first night following extubation are associated with sleep-disordered breathing. The secondary hypotheses are that duration of mechanical ventilation, BMI, and muscle strength are associated with sleep-disordered breathing during the night after extubation.

The secondary objective is to evaluate if sleep-disordered breathing in the ICU can be predicted by standard pulmonary function testing in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the SICU
2. Age over 18 years.
3. Ventilated patients with an endotracheal tube for at least 24 hours.

Exclusion Criteria:

1. Decreased level of consciousness as defined by a Richmond Agitation Sedation Scale (RASS) of 0.
2. Non-cooperative patient, CAM score positive for risk of delirium.
3. For women: pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ventilated patients in the surgical intensive unit (SICU)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 1 Night after extubation
  The apnea-hypopnea index (AHI) is calculated the night after extubation via a polysomnography device. An AHI ≥ 5 indicates sleep-disordered breathing and obstructive sleep apnea (OSA).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Mirzakhani H, Williams JN, Mello J, Joseph S, Meyer MJ, Waak K, Schmidt U, Kelly E, Eikermann M. Muscle weakness predicts pharyngeal dysfunction and symptomatic aspiration in long-term ventilated patients. Anesthesiology. 2013 Aug;119(2):389-97. doi: 10.1097/ALN.0b013e31829373fe. PMID 23584384
- [Derived] Timm FP, Zaremba S, Grabitz SD, Farhan HN, Zaremba S, Siliski E, Shin CH, Muse S, Friedrich S, Mojica JE, Kurth T, Ramachandran SK, Eikermann M. Effects of Opioids Given to Facilitate Mechanical Ventilation on Sleep Apnea After Extubation in the Intensive Care Unit. Sleep. 2018 Jan 1;41(1). doi: 10.1093/sleep/zsx191. PMID 29182729